CLINICAL TRIAL: NCT07377071
Title: Impact of Folate Administration on One-Year Mortality in Patients With Infection-Associated Acute Kidney Injury: An Open-Label Randomised Controlled Study
Brief Title: Folate Treatment to Reduce Death Risk in the Year After Infection-Related Acute Kidney Injury
Acronym: FOL-AKI
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Folate-AKI_HMRF2024
Record Dates: First submitted 2026-01-14; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-11

CONDITIONS: Infection-Associated Acute Kidney Injury
Keywords: Acute kidney injury; Cardiovascular events; Chronic kidney disease; Folate; Folic acid; Infection; Mortality; Open-label; Randomised controlled trial; Repurposing
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic; Infections | interventions — Folic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1. Usual care (No Intervention): Patients receive usual supportive management for infection-associated AKI (e.g., hemodynamic stabilization, fluid/electrolyte balance, antibiotics, cessation of nephrotoxic drugs, dialysis if needed), with no additional specific medication like folate.
- Arm 2. Folic acid 5 mg + Usual care (Experimental): Patients receive the same standard care as the control arm, plus folic acid (5 mg orally once daily, or via nasogastric tube if necessary) for a total duration of 90 days. Treatment starts immediately after randomization and recruitment.
  Interventions: Drug: Folic Acid 5 MG

INTERVENTIONS:
Drug: Folic Acid 5 MG — Oral folic acid 5 mg once daily for 90 days, administered as standard tablets (or via nasogastric tube if oral intake is not possible). Treatment is initiated immediately after randomization and diagnosis of infection-associated acute kidney injury (AKI per KDIGO criteria) and is given in addition to standard supportive AKI care. This low-dose regimen is selected based on preclinical evidence of oxidative stress reduction and Nrf2 activation in rat ischemia-reperfusion AKI models at low doses, and retrospective human data showing potential mortality benefit in infection-related AKI at similar oral doses (typically 5 mg daily). Duration of 90 days targets both acute recovery and early prevention of progression to chronic kidney disease (CKD). This differs from high-dose folic acid models (e.g., 250 mg/kg) used experimentally to induce AKI via crystal nephropathy, and from folate interventions in CKD or other populations.
  Other Names: Folate, Vitamin B9
  Arms: Arm 2. Folic acid 5 mg + Usual care

SUMMARY:
The goal of this clinical trial is to evaluate if taking folic acid (a form of vitamin B9) can help reduce the risk of death and improve kidney recovery in adults with acute kidney injury (AKI) caused by infections or sepsis.

The main question it aims to answer is: Does taking folic acid lower the chance of dying within one year for these patients? This study will also look at other important questions, such as whether folic acid helps kidneys recover faster (within 7 days), prevents long-term kidney problems (progression to chronic kidney disease at 3 months), reduces heart-related events, and is safe.

Researchers will compare the group receiving folic acid (5 mg taken by mouth once daily for 90 days, plus usual care) to the group receiving only usual care (standard treatments like fluids, blood pressure control, antibiotics, and stopping harmful medicines) to see if folic acid provides extra benefits.

Participants will:

1. Be randomly assigned to one of the two groups
2. Receive usual hospital care for their infection and AKI
3. Take the folic acid (or not, depending on their group) every day for 3 months
4. Have blood tests at the start and at 3 months (including to check serum folate levels)
5. Be followed up for 1 year through clinic visits, phone calls, or medical records to track health outcomes like survival, kidney function, and any side effects

This open-label study (both patients and doctors know which treatment is given) will include about 382 adults at Queen Mary Hospital in Hong Kong. It builds on earlier retrospective study data suggesting folic acid might improve survival in similar patients.

DETAILED DESCRIPTION:
1. Background Information Acute Kidney Injury (AKI) affects over 13 million people each year and has a hospital mortality of 20-40%. It is characterized by an abrupt loss of kidney function and is associated with multiple long-term sequelae including chronic kidney disease (CKD) and reliance on renal replacement therapy (RRT). Patients with AKI place a substantial financial burden on healthcare resources . Approximately 19%-37% of patients with AKI do not recover kidney function within one year, and 33% of patients progress to acute kidney disease (AKD), and from this subset, nearly 27% develop CKD within 90 days post-AKI diagnosis. This highlights the critical importance of early detection and effective management of AKI to prevent progression.

   1.1 Epidemiology of AKI AKI affects all countries, and its prevalence ranges from <1% to 66%. Apart from population variation, different classification systems used in epidemiological studies contributes to the varied estimation of AKI incidence. Little epidemiological data is available for AKI in Hong Kong (HK). Szeto and Pang reported AKI was present in 9.1% of all adult hospital admissions in HK. The crude mortality rate of AKI in patients attending an emergency department (ED) in HK is 25%.

   1.2 Etiology of AKI AKI is a complex syndrome. The causes of AKI can be classified into prerenal, intrinsic renal and postrenal. Prerenal causes involve reduced renal perfusion due to medications, heart failure, infections, sepsis or volume depletion (e.g., diuretic overuse, severe dehydration and diarrhea). Intrinsic renal causes involve direct damage to the kidney structures including pre-existing renal impairment (e.g., glomerulonephritis, interstitial nephritis and vasculitis), and nephrotoxic drugs. Postrenal AKI is due to obstruction of urinary flow (e.g., kidney stone and tumors), and is especially common in elderly men. Sepsis, infections and use of nephrotoxic drugs are common causes of AKI overall, leading to reduced renal blood flow. In intensive care unit (ICU) settings, AKI occurs in more than half of patients, and half of all patients with AKI in ICU have sepsis. Drug induced AKI occurs in 20% of hospital cases. Associated drugs include non-steroidal anti-inflammatory drugs (NSAIDs), angiotensin converting enzyme inhibitors (ACEI), angiotensin II receptor blockers [ARBs], metformin, aminoglycosides, diuretics and iodine containing X-ray contrast.

   The diverse etiologies of AKI along with other comorbidities make it difficult to determine and understand the pathophysiology of AKI. Recently, oxidative stress has been accepted as the primary mediator of adverse outcomes in AKI, playing a critical role in both initiating and further development of AKI. In the context of deficient renal blood flow in AKI, ischemia-reperfusion represents the most common mechanism in which oxygen and nutrient delivery as well as waste removal are impaired; this mismatch of oxygen supply and demand, and accumulation of waste lead to cellular injury and even death. Sepsis-induced AKI also triggers oxidative stress. Oxidative stress as a key component in the pathophysiology of AKI provides a target for potential therapeutics.

   1.3 Treatment for AKI The KDIGO serum creatinine-based criteria is mostly used to stage AKI. The management of AKI is primarily supportive. The key to management is assuring hemodynamic stability and preventing hypovolemia so as to ensure sufficient renal perfusion. Depending on the cause and severity of AKI, treatments in hospital usually include: blood pressure and circulating electrolyte control; body fluid balance (e.g., with fluid replacement and/or diuretics); review and cessation of nephrotoxic medication; removing the obstruction if there is obstruction; and use of antibiotics. Malnutrition also affects patients with AKI, which requires a kidney-friendly diet, adequate nutrition and restricting potassium. There are no approved pharmacological agents for treating AKI.

   1.4 Folate Folate (vitamin B9) occurs naturally in foods. Folic acid is a synthetic, parent compound of folate family. Folic acid gets metabolized into 5-methyltetrahydrofolate (5-MTHF). 5-MTHF is the biologically active form of folate and the predominant form of dietary folate in plasma.

   A systematic review was conducted in accordance with the PRISMA guidelines and registered in PROSPERO (CRD42024589377). The investigators searched six databases (PubMed, MEDLINE, CINAHL, CENTRAL, Embase, and Web of Science) from their inception until March 2024, identifying 36 randomized controlled trials (RCTs) that evaluated folate use in patients with CKD or AKI. Of these, 22 RCTs compared folate use with no use in patients with CKD, with treatment durations ranging from 4 weeks to 4.5 median years, and majority use folic acid. Notably, no published data focused on AKI populations. Among included RCTs, 20 reported that folate use significantly reduced homocysteine (Hcy) levels but not directly reduced cardiovascular events in CKD patients. Only 5 trials assessed markers of kidney disease progression including 3 measured serum creatinine and 2 measured estimated glomerular filtration rate (eGFR) with inconsistent findings. The largest study, China Stroke Primary Prevention Trial with 1671 CKD patients, demonstrated that folate use slowed the annual decline in eGFR compared to controls (0.96 ± 5.81% vs. 1.72 ± 6.08%, respectively). Similarly, Chang et al. observed a modest reduction in serum creatinine in end-stage renal disease (ESRD) patients receiving folate (10.94 ± 2.01 vs. 11.30 ± 2.31 in controls). Safety analyses across all 22 RCTs revealed no severe adverse events attributable to folate, and no significant differences in adverse outcomes were noted between the treatment and control groups.

   Low doses: In a rat model of AKI with ischemia-reperfusion, 5-MTHF at a low dose of 3 μg/kg body weight improved kidney function, reduced plasma creatinine levels and alleviate oxidative stress within 24 hours. The expression of neutrophil gelatinase-associated lipocalin (NGAL), a marker of proximal tubular injury, was significantly reduced after folate treatment. 5-MTHF activated the nuclear factor erythroid 2-related factor 2 (Nrf2), a key regulator of the antioxidant defense system. Nrf2 activation regulates gene expression of detoxification enzymes and antioxidant proteins, which is vital to restore antioxidant defense against oxidative stress injury. Oxidative stress is the mainstay responsible to the adverse outcomes in AKI. The expression of antioxidant enzymes, superoxide dismutase-1 (SOD-1), glutathione synthesizing enzymes and heme oxygenase-1 (HO-1), were all upregulated after folate treatment.

   High doses: Folic acid, a precursor of folate, at high doses, e.g., 250 mg/ /kg body weight, is used to induce AKI in animals. High doses of folic acid remain unmetabolized and cause AKI due to the rapid onset of folic acid crystals within renal tubules with a consequent acute tubular necrosis, epithelial regeneration and renal cortical scarring. This is only experimental in animals, and high levels of folic acid have not been observed in the clinic kidney diseases.

   Preliminary data The investigators conducted a retrospective study to characterize the epidemiology and outcomes of adult patients with presumed infections and diagnosed with AKI at Queen Mary Hospital (QMH). The study utilized data from the Clinical Data Analysis and Reporting System (CDARS) of the Hospital Authority (HA) for the period between January 1, 2023, and December 31, 2023. Inclusion criteria required patients to be aged 18 years or older, have an infection, and be diagnosed with AKI based on the Kidney Disease: Improving Global Outcomes (KDIGO) criteria. A total of 2585 patients met the eligibility criteria, with a median age of 72 [IQR: 61, 84] years and 56.0% being male. The median length of hospital stay was 13 [IQR: 6, 26] days. Notably, 61.2% (1581 patients) recovered quickly within one day, and by 7 days 23.4% (605 patients) did not recover and majority of them (543 patients) remained unrecovered by 28 days. 28.1% (727 patients) had sepsis, and 13.8% (357 patients) had pre-existing CKD. Among patients without pre-existing CKD, 1.5% (33 patients) developed CKD at 3 months post AKI diagnosis. The one-year mortality was 23.2% (600 patients).

   A retrospective analysis comparing folic acid users (206 patients) and non-users (2379 patients) was conducted. Folic acid was prescribed at the same time when AKI occurred. Majority (178 patients) received an oral dose of 5 mg folic acid daily. The median treatment period was 35.5 days [IQR 13.25, 83]. Results revealed that folic acid users had slightly higher rates of AKI recovery at 24 hours (64.1% vs. 60.9%) and 7 days (79.1% vs. 76.4%), and had a significantly lower one-year mortality [11.6% vs. 24.2% (24 vs. 576 patients), P < 0.001], compared with non-users. The progression to CKD at 3 months and cardiovascular events over one year post AKI showed no significant differences. The investigators conducted a multivariate logistic regression analysis to analyze the confounding factors including age, gender, CKD, diabetes mellitus, hypertension, heart failure, ischemic heart disease, stroke and sepsis, and confirmed the use of folic acid contributed to 57% [OR 0.428 (95% CI: 0.275, 0.666), P = 0.0002] of reducing mortality risk. Age, stroke and sepsis increased mortality risk; gender, diabetes mellitus, hypertension, heart failure, and ischemic heart disease did not significantly affect patient mortality; and CKD unexpectedly decreased mortality risk by 28% (P= 0.0325). Patients with CKD are often under more intense medical surveillance and management, and receive more comprehensive care, which may contribute to better overall health and increased survival.

   The discrepancy between one-year mortality reduction and non-significant AKI recovery may reflect the multifactorial nature of mortality in AKI patients. While early renal recovery is important, long-term survival is influenced by systemic inflammation, cardiovascular events, and nutritional status. Folate's known roles in endothelial function, homocysteine metabolism, and oxidative stress modulation may confer survival benefits independent of short-term renal recovery.

   The investigators hypothesize that the observed mortality reduction is mediated by mechanisms beyond immediate renal function improvement. Sepsis, the leading cause of AKI in critically ill patients, triggers a systematic inflammatory response and a surge in reactive oxygen species that cause widespread cellular damage. Folate has been shown to alleviate oxidative stress in a rat model of AKI. Folate's benefit may lie in attenuating systemic oxidative stress. Moreover, AKI recovery defined by serum creatinine has inherent limitations. Creatinine is a delayed and imperfect marker of kidney function, especially in sepsis. Septic AKI involves complex pathophysiology including tubular injury, microvascular dysfunction, and systemic inflammation, which is not adequately represented by creatinine levels alone. A prospective randomized controlled trial is important to confirm or refute the observation, and to investigate the causal link between folate and improved survival.

   To further explore the influence of CKD status, subgroup analyses were conducted. Among 357 patients with CKD, folic acid users (n = 55) had relatively higher AKI recovery rates at 24 hours (74.5% vs. 73.2%), 7 days (87.3% vs. 84.4%), and 28 days (89.1% vs. 85.1%), along with significantly lower one-year mortality (5.5% vs. 20.5%, P = 0.0069). In the cohort without CKD (n = 2228), folic acid users (n = 151) had comparable AKI recovery rates to non-users at 24 hours (62.9% vs. 61.8%), 7 days (78.8% vs. 79.0%), and 28 days (78.8% vs. 79.8%), and still showed significantly lower one-year mortality (13.9% vs. 24.7%, P = 0.0021). Compared to the overall cohort, subgroup analyses revealed a consistent trend of reduced one-year mortality among folic acid users, regardless of CKD status.

   These findings suggest folate has potential to improve AKI recovery and decrease patient mortality, warranting further investigation in the proposed study. The retrospective study, however, is limited by the cohort selection which was not rigorously matched between treatment and control groups, and the period of folate treatment varied. There might be unidentified confounding factors and selection bias of folic acid effect on mortality. Therefore, there is a compelling need to conduct a thorough clinical study to investigate the role of folate administration on AKI patient outcomes.

   1.5 Unmet Clinical Need AKI is a common health issue with high morbidity and mortality in hospital. Delays in detection and treatment result in an in-hospital mortality rate of 20-40% that is higher than acute stroke and acute myocardial infarction combined. Management of AKI is primarily supportive. There are no approved pharmacological agents for treating AKI. Oxidative stress provides a target for therapeutics. Animal experiments have shown folate IN LOW DOSES alleviated oxidative stress, decreased plasma creatinine levels and improved kidney function of AKI. Folate administration has been studied to improve survival of patients with CKD using randomized clinical trials. Evidence for the protective effect of folate against AKI to safely reduce circulating creatinine levels, progression to CKD/ESRD and mortality in adult patients with AKI is needed.

   1.6 Impact If folate treatment improved outcome for 1% cases, as the global burden of AKI per year is 13 million cases, then potentially 130,000 patients could benefit per year; in HK, as AKI identiﬁed with a crude hospital admission of 12%, among around 2 million hospital admissions in one year, potentially 2,500 patients could benefit per year.
2. Aims and Hypotheses 2.1 Aims This study aims to test folate administration in adult patients with an infection experiencing AKI for the effectiveness on mortality and kidney function recovery.

2.2 Hypothesis The hypothesis of this study is that folate administration plus standard care will reduce mortality and improve kidney function recovery, compared to standard care alone.

2.3 Objectives

1. To assess how effective folate administration is on reducing the one-year mortality
2. To assess how effective folate administration is on improving AKI recovery within 7 days, and preventing the progression to CKD at 3 months
3. To assess how effective folate administration is on reducing cardiovascular events over the study period

3 Plan of Investigation 3.1 Subjects In order to reduce variability and confounding factors introduced by diverse etiologies of AKI, the investigators focus on AKI associated with infections including sepsis.

3.1.1 Inclusion criteria

Patients will be eligible for the study if ALL the following are present:

1. Adults ≥18 years of age;
2. Presence of an infection;
3. Diagnosed with AKI based on KDIGO criteria;
4. Ability to provide informed consent or having a legally authorized representative to provide consent.

3.1.2 Exclusion criteria

Patients will be excluded from the study if any of the following conditions is present:

1. Patients with AKI due to causes not infections or sepsis (e.g., nephrotoxic drugs or obstruction of urinary flow);
2. Known hypersensitivity or contraindication to folate;
3. Pregnancy or breastfeeding women;
4. Already on folate treatment

3.1.3 Sample Size From the retrospective study of AKI patients at QMH from CDARS, folic acid non-users have 76.4% AKI recovery (23.6% non-recovery) at 7 days, and 24.2% one-year mortality. Folic acid users have 20.9% non-recovery at 7 days, and 11.6% one-year mortality.

If the investigators assume that folate administration plus standard care reduces one-year mortality from 24.2% to 11.6%, 191 participants per group will be needed to detect a significant difference with 90% power at the 5% level. Thus, the total sample size would be 382 participants.

For AKI recovery, the number of patients (9968) required to detect a significant difference with 90% power at the 5% level will be too many to be handled in this study. Also, the patient availability is limited in the single-center design considering there were 2585 patients identified in QMH in 2023.

3.2 Methods 3.2.1 Study design An open-label, randomized controlled trial with 1:1 ratio.

Arm 1. Control group (no specific medication) Arm 2. Folate group (5 mg folic acid, taken orally once daily for 90 days)

All patients diagnosed with AKI will receive standard care. The medications will be initiated right after AKI patients are recruited.

Follow-up visits: At 3 and 12 months.

This study will be conducted in compliance with the principles of the Declaration of Helsinki and the International Council for Harmonization Guideline for Good Clinical Practice (ICH-GCP, ICH E6[R3]) and reported in accordance with the Consolidated Standards of Reporting Trials (CONSORT) statement.

3.2.2 Screening, recruitment and consent First, the investigators will check hospital records and the Clinical Management System (CMS) to identify potential participants. Second, the investigators will use a screening form to determine the eligibility of potential participants, and review their medical records. Third, the investigators will access eligible patients to inform the study and ask for their consent to participate.

3.2.3 Randomization To ensure balanced allocation across treatment arms and address potential confounding due to pre-existing CKD, stratified block randomization will be employed. Patients will be stratified by CKD status (presence vs. absence) prior to randomization. Within each stratum, block randomization will be conducted to assign participants to either the control group or the 5 mg/day folic acid group.

An investigator with no clinical involvement in the trial will do block randomization using www.randomization.com. Separate randomization lists will be created for CKD and non-CKD strata to maintain balance across arms. He/she will keep the original random allocation sequences in an inaccessible third place and works with a copy.

The study information and medications will be put into sealed envelopes. The outside of the envelope will contain the name of the study and possible arms contained within, but not which arm is selected. Each enrolled patient will be assigned an order number and receive the corresponding envelope. The patient ID, date, time and other information will be recorded on the envelope. Once the patients completed all baseline assessments, the patients will be allocated the treatment. In the case of broken or lost envelopes, the researcher figures out what the number of the envelope it is and replaces the envelope with the same treatment according to the allocation.

3.2.4 Usual care Depending on the cause and severity of AKI, usual care in hospital includes: blood pressure and circulating electrolyte control; body fluid balance (e.g., with fluid replacement and/or diuretics); review and cessation of nephrotoxic medication; removing the obstruction if there's a blockage; and use of antibiotics. In severe cases, dialysis may be needed. Usual care is according to physician acumen and clinical story.

3.2.5 Data collection The investigators will collect data and follow-up assessments. The baseline data includes demographics, medical history, medication use, physical examination, diagnostics, kidney function parameters, nutrition histology, and standard care received. Serum folate levels will be measured at baseline and at 3 months. The follow-up scheduled at 3 and 12 months includes visit information, clinical outcomes, kidney function parameters, and any adverse events. Follow-up will include in-person visits, telephone calls, telehealth consultations, and electronic health record review.

The investigators will monitor patient adherence by regular follow-up calls and check-ins, and encourage adherence. The investigators will address safety concerns and issues promptly.

The data will be collected into an IT system that requires a password to access, and only authorized personnel can access. The data will be entered in real time, and the database will be regularly checked to ensure accuracy and completeness. All study staff involved in data collection will get trained rigorously to ensure confidentiality, integrity and availability of the database.

3.2.6 Study Sites This study will be conducted at one hub hospital (Local Clinical Centre (LCC), QMH) within HK. Patients will be recruited from the ED, wards and ICU with subsequent follow-up in the medical wards, ICUs and home (when discharged). At the LCC, a lead investigator will be responsible for study activities but much of the work will be carried out by medical staff attending patients with AKI within the hospital and by hospital and university research nurses.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for the study if ALL the following are present:

1. Adults ≥18 years of age
2. Presence of an infection (defined by clinical signs/symptoms such as fever, chills, or laboratory evidence; or presumed infection indicated by blood culture obtained and at least 4 Qualifying Antimicrobial Days starting within 2 calendar days before/after blood culture; or physician's judgment)
3. Diagnosed with AKI based on KDIGO criteria: increase in serum creatinine by ≥0.3 mg/dL (26.5 µmol/L) within 48 hours, OR increase to ≥1.5 times baseline, OR urine output <0.5 mL/kg/h for ≥6 hours (baseline creatinine is the median from 8-365 days prior, or lowest from 0-7 days if unavailable)
4. Ability to provide informed consent or having a legally authorized representative to provide consent

Exclusion Criteria:

Patients will be excluded from the study if any of the following conditions is present.

1. Patients with AKI due to causes not related to infections or sepsis (e.g., nephrotoxic drugs, obstruction of urinary flow)
2. Known hypersensitivity or contraindication to folate (folic acid)
3. Pregnancy or breastfeeding women
4. Already on folate treatment at the time of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
All-Cause Mortality at 1 Year | Up to 365 days (1 year) from randomization
  The proportion of participants who die from any cause within 1 year after randomization. Mortality will be determined from hospital records, follow-up visits, telephone calls, or electronic health records. Events will be adjudicated if needed.

SECONDARY OUTCOMES:
AKI Recovery Rate at 7 Days | 7 days after randomization
  The proportion of participants who achieve AKI recovery within 7 days after randomization, defined as alive and no longer meeting KDIGO criteria for even Stage 1 AKI (return to baseline creatinine or below Stage 1 threshold), or as per treating physician judgment.
Progression to Chronic Kidney Disease (CKD) at 3 Months | 3 months (90 days) after randomization
  In participants without pre-existing CKD at baseline, the proportion who develop CKD (defined by KDIGO criteria, e.g., persistent eGFR <60 mL/min/1.73m² or other markers) at 3 months post-randomization.
Incidence of Major Adverse Cardiovascular Events (MACE) at 1 Year | Up to 365 days from randomization
  The proportion of participants experiencing MACE (composite of acute myocardial infarction, stroke, cardiovascular death, acute coronary syndrome/ischemic heart disease, or heart failure) over 1 year. Events will be adjudicated by a blinded clinical endpoint committee (senior clinicians from Emergency Medicine, Nephrology, and Cardiology).
Incidence of Adverse Events | Up to 365 days from randomization
  The number and proportion of participants experiencing adverse events (including serious adverse events), classified by nature, intensity, duration, and causality to study treatment (folic acid). Safety monitoring per protocol.
Serum Folate Levels Comparison | Baseline and 3 months after randomization
  Comparison of serum folate levels between groups and correlation with outcomes (e.g., low vs. high levels at baseline and 3 months)
Change in Serum Creatinine | Baseline, up to 30 days from randomization, 3 months after randomization, and 1 year after randomization
  Change in serum creatinine levels (in µmol/L or mg/dL) from baseline to specified time points during hospitalization and follow-up. Measured via standard laboratory assays.
Change in Estimated Glomerular Filtration Rate (eGFR) | Baseline, up to 30 days from randomization, 3 months after randomization, and 1 year after randomization
  Change in eGFR (calculated using standard equations, e.g., CKD-EPI) from baseline to key time points during hospital stay and follow-up.
Change in Urine Output | Up to 30 days from randomization
  Daily or cumulative urine output (in mL/kg/h or total mL) monitored via indwelling catheter or timed collections where clinically indicated
Change in Blood Urea Nitrogen (BUN) | Baseline, up to 30 days from randomization, 3 months after randomization, and 1 year after randomization
  Change in blood urea nitrogen levels (in mmol/L or mg/dL) from baseline. Measured via standard laboratory assays.
Incidence of Proteinuria | Up to 30 days from randomization and at 3 months after randomization
  Proportion of participants with new or worsening proteinuria (e.g., urine protein-to-creatinine ratio >0.3 g/g or dipstick ≥1+).
Time to AKI Recovery | Up to 30 days from randomization
  Time (in days) from randomization to AKI recovery, defined as alive and no longer meeting KDIGO criteria for even Stage 1 AKI (return of serum creatinine to baseline or below Stage 1 threshold, or per treating physician judgment). Assessed daily during hospitalization.
Incidence of Renal Replacement Therapy (RRT) Initiation | Up to 90 days from randomization
  Proportion of participants requiring initiation of any form of renal replacement therapy (e.g., intermittent hemodialysis, continuous venovenous hemofiltration).
Duration of Renal Replacement Therapy | Up to 90 days from randomization
  Total duration (in days) of renal replacement therapy among participants who receive it.
Hospital Length of Stay | Up to 90 days from randomization
  Total duration of hospitalization (in days) from randomization to discharge.
Intensive Care Unit (ICU) Length of Stay | Up to 90 days from randomization
  Total duration of ICU stay (in days) from randomization among participants admitted to ICU.
Incidence of Hospital Readmissions Due to Kidney-Related Issues | Up to 365 days from randomization
  Proportion of participants with hospital readmissions primarily due to kidney-related complications (e.g., worsening renal function, fluid overload, electrolyte imbalance). Adjudicated from medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Yaqing Jiao, PhD, Principal Investigator — Department of Emergency Medicine, The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No